CLINICAL TRIAL: NCT06357923
Title: Study of the Evolution of the Expression of the LAMP-2 Protein During the Advance as Well as Variations and Allelic Mutations in the Main Genes Involved in the Occurrence of Age-related Myelodysplastic Syndromes
Brief Title: Study of the Evolution of the Expression of the LAMP-2 Protein During the Advance in Age
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 23-PP-13; 2024-A00321-46 (Other: ANSM)
Record Dates: First submitted 2024-04-05; First posted 2024-04-10 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-09

CONDITIONS: Aging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- evaluation of LAMP-2 protein expression (Other): dosing of level expression of LAMP-2
  Interventions: Diagnostic Test: dosage

INTERVENTIONS:
Diagnostic Test: dosage — Presence of mutation on the gene panel and Frequency of allele variation

SUMMARY:
Recruitment on the RAV pole in consultation or day hospital. Competitive recruitment of subjects > 60 years of age respecting a male/female ratio = 1.

DETAILED DESCRIPTION:
Recruitment on the RAV pole in consultation or day hospital. Competitive recruitment of subjects > 60 years of age respecting a male/female ratio = 1. After explanations and collection consent, collection of the patient's socio-demographic and medical characteristics and then carrying out a Peripheral venous blood sample (2 x 5ml tubes).

ELIGIBILITY:
Inclusion Criteria:

* Men and women over 60 years of age.

Exclusion Criteria:

* Inability to Understand Consent,
* Non-Security Beneficiaries
* social, subjects protected by law, subjects deprived of liberty,
* history of breast cancer,
* brain tumor,
* melanoma,
* colon cancer,
* lung cancer,
* prostate cancer,
* lymphoma,
* myeloma,
* syndrome myelodysplastic/myeloproliferative,
* leukemia,
* history of radiation therapy.

Ages: 60 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-09-26 (Actual); Primary Completion 2026-09-26 (Estimated); Study Completion 2026-09-26 (Estimated)

PRIMARY OUTCOMES:
Expression level of LAMP2 (protein and isoform A and B mRNA) | day 0
  dosage

SECONDARY OUTCOMES:
Presence of mutation in the "Oncomin Myeloid Reasearch Assay" gene panel targeting approximately 40 Different genes | day 0
  dosage

CONTACTS AND LOCATIONS:
Overall Officials: Andrea CICCONE, Principal Investigator — Centre Hospitalier Universitaire de Nice
Locations (1):
- Chu de Nice, Nice, France

IPD SHARING:
Plan to Share IPD: No